CLINICAL TRIAL: NCT01927354
Title: Observational Study on the Investigation of the Molecular Mechanism and Clinical Significance of the Interplay Between Twist1 and Other EMT Regulators Through microRNA-29 Family.
Brief Title: Study on the Interplay Between Twist1 and Other EMT Regulators Through microRNA-29 Family.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201112085RID
Record Dates: First submitted 2013-08-07; First posted 2013-08-22 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2013-09

CONDITIONS: Head-and-Neck Squamous Cell Carcinoma
Keywords: Head-and-Neck squamous cell carcinoma (HNSCC); epithelial-mesenchymal transition (EMT); microRNA29; Twist1
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Acrocephalosyndactylia

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples With DNA — tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Head and neck cancer: Subjects who suffer from oral cancer. Collect a 0.5x0.5Cm2 tissue sample of the tumor during the surgery.

SUMMARY:
Investigation of the molecular mechanism and clinical significance of the interplay between Twist1 and other EMT regulators through microRNA-29 family.

DETAILED DESCRIPTION:
Head and neck squamous cell carcinoma (HNSCC) is one of the leading causes of cancer deaths worldwide, and it ranks the fourth male cancer-related death in Taiwan. In HNSCC, invasiveness and metastasis of cancer cells contribute to the major cause of mortality; therefore, elucidation of the mechanism and development of new strategies against metastasis is the utmost importance in treating advanced HNSCC. Epithelial-mesenchymal transition (EMT) is a process by which epithelial cells lose their polarity and are converted to a mesenchymal phenotype, and recently is considered as the major mechanism for cancer metastasis. The initiation of EMT is hallmarked by suppression of the intercellular junctional protein E-cadherin by a variety of transcriptional factors, including Twist1, Snail, Slug, SIP1, Zeb1 and E47. However, during metastatic evolution, the interplay between different EMT inducers has been investigated limitedly. Previously study demonstrated that hypoxia induces EMT of HNSCC through induction of Twist1 expression. Additionally showed that Twist1 promotes EMT and tumor-initiating capability through upregulation of Bmi1, and co-expression Twist1 and Bmi1 predicts a worse prognosis of HNSCC cases. Accumulated evidence suggests that microRNAs play essential roles in cancer progression and metastasis. Therefore, we aim to investigate the role of microRNA in Twist1-mediated cancer metastasis, and the interplay between Twist1 and other EMT regulators. Our preliminary data showed that the expression of miR-29 family, including miR-29a, b, and c were increased in Twist1-overexpressing HNSCC cells. Furthermore, we discovered that SIN3A, a co-repressor of another EMT regulator Snail, is a target of miR-29s. We therefore speculate that Twist1 modifies the function of Snail through microRNA machinery. In this proposal, we will delineate the regulatory mechanism of the Twist1-miR29s-SIN3A axis. We will also investigate the molecular interplay between Twist1 and Snail through Twist1-miR29s-SIN3A signal pathway. Furthermore, we will elucidate the molecular basis and pathophysiologic significance of Twist1-Snail interaction under hypoxic environment. Finally, we will confirm the in vitro finding by in vivo animal study and HNSCC samples. These results will provide crucial information for understanding the molecular basis of HNSCC metastasis, and will be valuable for developing new therapeutic strategies against advanced HNSCC.

ELIGIBILITY:
Inclusion Criteria:

* Head and neck cancer

Exclusion Criteria:

* pregnant woman

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Medical center
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
The interplay between Twist1 and other EMT regulators throigh microRNA-29 family | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Shin-Jung Cheng, DDS, MS, PhD, Principal Investigator
Locations (1):
- National Taiwan University Hospital research Ethics Committee, Taipei, Taiwan

REFERENCES:
- [Background] Department of health, the Executive Yuan, R.O.C. Cancer Registry Annual Report in Taiwan area, 2007. Goldenberg D, Lee J, Koch WM, et al.
- [Background] Goldenberg D, Lee J, Koch WM, Kim MM, Trink B, Sidransky D, Moon CS. Habitual risk factors for head and neck cancer. Otolaryngol Head Neck Surg. 2004 Dec;131(6):986-93. doi: 10.1016/j.otohns.2004.02.035. PMID 15577802
- [Background] Haffty BG. Concurrent chemoradiation in the treatment of head and neck cancer. Hematol Oncol Clin North Am. 1999 Aug;13(4):719-42, vi-vii. doi: 10.1016/s0889-8588(05)70088-5. PMID 10494509
- [Background] Gilbert J, Forastiere AA. Organ preservation trials for laryngeal cancer. Otolaryngol Clin North Am. 2002 Oct;35(5):1035-54, vi. doi: 10.1016/s0030-6665(02)00035-x. PMID 12587246
- [Background] Fanucchi M, Khuri FR. Chemotherapy for recurrent or metastatic squamous cell carcinoma of the head and neck. Semin Oncol. 2004 Dec;31(6):809-15. doi: 10.1053/j.seminoncol.2004.09.014. PMID 15599859
- [Background] Papadimitrakopoulou VA, Izzo J, Mao L, Keck J, Hamilton D, Shin DM, El-Naggar A, den Hollander P, Liu D, Hittelman WN, Hong WK. Cyclin D1 and p16 alterations in advanced premalignant lesions of the upper aerodigestive tract: role in response to chemoprevention and cancer development. Clin Cancer Res. 2001 Oct;7(10):3127-34. PMID 11595705
- [Background] Farrar M, Sandison A, Peston D, Gailani M. Immunocytochemical analysis of AE1/AE3, CK 14, Ki-67 and p53 expression in benign, premalignant and malignant oral tissue to establish putative markers for progression of oral carcinoma. Br J Biomed Sci. 2004;61(3):117-24. doi: 10.1080/09674845.2004.11732655. PMID 15462255
- [Background] Gold KA, Lee HY, Kim ES. Targeted therapies in squamous cell carcinoma of the head and neck. Cancer. 2009 Mar 1;115(5):922-35. doi: 10.1002/cncr.24123. PMID 19156911
- [Background] Nathan CO, Amirghahari N, Abreo F, Rong X, Caldito G, Jones ML, Zhou H, Smith M, Kimberly D, Glass J. Overexpressed eIF4E is functionally active in surgical margins of head and neck cancer patients via activation of the Akt/mammalian target of rapamycin pathway. Clin Cancer Res. 2004 Sep 1;10(17):5820-7. doi: 10.1158/1078-0432.CCR-03-0483. PMID 15355912
- [Background] Nakayama H, Ikebe T, Beppu M, Shirasuna K. High expression levels of nuclear factor kappaB, IkappaB kinase alpha and Akt kinase in squamous cell carcinoma of the oral cavity. Cancer. 2001 Dec 15;92(12):3037-44. doi: 10.1002/1097-0142(20011215)92:123.0.co;2-#. PMID 11753981
- [Background] Thiery JP. Epithelial-mesenchymal transitions in tumour progression. Nat Rev Cancer. 2002 Jun;2(6):442-54. doi: 10.1038/nrc822. No abstract available. PMID 12189386
- [Background] Higgins DF, Kimura K, Bernhardt WM, Shrimanker N, Akai Y, Hohenstein B, Saito Y, Johnson RS, Kretzler M, Cohen CD, Eckardt KU, Iwano M, Haase VH. Hypoxia promotes fibrogenesis in vivo via HIF-1 stimulation of epithelial-to-mesenchymal transition. J Clin Invest. 2007 Dec;117(12):3810-20. doi: 10.1172/JCI30487. PMID 18037992
- [Background] Thompson EW, Newgreen DF, Tarin D. Carcinoma invasion and metastasis: a role for epithelial-mesenchymal transition? Cancer Res. 2005 Jul 15;65(14):5991-5; discussion 5995. doi: 10.1158/0008-5472.CAN-05-0616. No abstract available. PMID 16024595
- [Background] Thiery JP, Sleeman JP. Complex networks orchestrate epithelial-mesenchymal transitions. Nat Rev Mol Cell Biol. 2006 Feb;7(2):131-42. doi: 10.1038/nrm1835. PMID 16493418
- [Background] Tamura G, Yin J, Wang S, Fleisher AS, Zou T, Abraham JM, Kong D, Smolinski KN, Wilson KT, James SP, Silverberg SG, Nishizuka S, Terashima M, Motoyama T, Meltzer SJ. E-Cadherin gene promoter hypermethylation in primary human gastric carcinomas. J Natl Cancer Inst. 2000 Apr 5;92(7):569-73. doi: 10.1093/jnci/92.7.569. PMID 10749913
- [Background] Peinado H, Ballestar E, Esteller M, Cano A. Snail mediates E-cadherin repression by the recruitment of the Sin3A/histone deacetylase 1 (HDAC1)/HDAC2 complex. Mol Cell Biol. 2004 Jan;24(1):306-19. doi: 10.1128/MCB.24.1.306-319.2004. PMID 14673164
- [Background] Blanco MJ, Moreno-Bueno G, Sarrio D, Locascio A, Cano A, Palacios J, Nieto MA. Correlation of Snail expression with histological grade and lymph node status in breast carcinomas. Oncogene. 2002 May 9;21(20):3241-6. doi: 10.1038/sj.onc.1205416. PMID 12082640
- [Background] Elloul S, Elstrand MB, Nesland JM, Trope CG, Kvalheim G, Goldberg I, Reich R, Davidson B. Snail, Slug, and Smad-interacting protein 1 as novel parameters of disease aggressiveness in metastatic ovarian and breast carcinoma. Cancer. 2005 Apr 15;103(8):1631-43. doi: 10.1002/cncr.20946. PMID 15742334
- [Background] Shih JY, Tsai MF, Chang TH, Chang YL, Yuan A, Yu CJ, Lin SB, Liou GY, Lee ML, Chen JJ, Hong TM, Yang SC, Su JL, Lee YC, Yang PC. Transcription repressor slug promotes carcinoma invasion and predicts outcome of patients with lung adenocarcinoma. Clin Cancer Res. 2005 Nov 15;11(22):8070-8. doi: 10.1158/1078-0432.CCR-05-0687. PMID 16299238
- [Background] Rosivatz E, Becker I, Specht K, Fricke E, Luber B, Busch R, Hofler H, Becker KF. Differential expression of the epithelial-mesenchymal transition regulators snail, SIP1, and twist in gastric cancer. Am J Pathol. 2002 Nov;161(5):1881-91. doi: 10.1016/S0002-9440(10)64464-1. PMID 12414534
- [Background] Pena C, Garcia JM, Garcia V, Silva J, Dominguez G, Rodriguez R, Maximiano C, Garcia de Herreros A, Munoz A, Bonilla F. The expression levels of the transcriptional regulators p300 and CtBP modulate the correlations between SNAIL, ZEB1, E-cadherin and vitamin D receptor in human colon carcinomas. Int J Cancer. 2006 Nov 1;119(9):2098-104. doi: 10.1002/ijc.22083. PMID 16804902
- [Background] Gupta GP, Massague J. Cancer metastasis: building a framework. Cell. 2006 Nov 17;127(4):679-95. doi: 10.1016/j.cell.2006.11.001. PMID 17110329
- [Background] Harris AL. Hypoxia--a key regulatory factor in tumour growth. Nat Rev Cancer. 2002 Jan;2(1):38-47. doi: 10.1038/nrc704. PMID 11902584
- [Background] Semenza GL. HIF-1 and tumor progression: pathophysiology and therapeutics. Trends Mol Med. 2002;8(4 Suppl):S62-7. doi: 10.1016/s1471-4914(02)02317-1. PMID 11927290
- [Background] Peinado H, Olmeda D, Cano A. Snail, Zeb and bHLH factors in tumour progression: an alliance against the epithelial phenotype? Nat Rev Cancer. 2007 Jun;7(6):415-28. doi: 10.1038/nrc2131. Epub 2007 May 17. PMID 17508028
- [Background] Imai T, Horiuchi A, Wang C, Oka K, Ohira S, Nikaido T, Konishi I. Hypoxia attenuates the expression of E-cadherin via up-regulation of SNAIL in ovarian carcinoma cells. Am J Pathol. 2003 Oct;163(4):1437-47. doi: 10.1016/S0002-9440(10)63501-8. PMID 14507651
- [Background] Krishnamachary B, Zagzag D, Nagasawa H, Rainey K, Okuyama H, Baek JH, Semenza GL. Hypoxia-inducible factor-1-dependent repression of E-cadherin in von Hippel-Lindau tumor suppressor-null renal cell carcinoma mediated by TCF3, ZFHX1A, and ZFHX1B. Cancer Res. 2006 Mar 1;66(5):2725-31. doi: 10.1158/0008-5472.CAN-05-3719. PMID 16510593
- [Background] Evans AJ, Russell RC, Roche O, Burry TN, Fish JE, Chow VW, Kim WY, Saravanan A, Maynard MA, Gervais ML, Sufan RI, Roberts AM, Wilson LA, Betten M, Vandewalle C, Berx G, Marsden PA, Irwin MS, Teh BT, Jewett MA, Ohh M. VHL promotes E2 box-dependent E-cadherin transcription by HIF-mediated regulation of SIP1 and snail. Mol Cell Biol. 2007 Jan;27(1):157-69. doi: 10.1128/MCB.00892-06. Epub 2006 Oct 23. PMID 17060462
- [Background] Ip YT, Park RE, Kosman D, Yazdanbakhsh K, Levine M. dorsal-twist interactions establish snail expression in the presumptive mesoderm of the Drosophila embryo. Genes Dev. 1992 Aug;6(8):1518-30. doi: 10.1101/gad.6.8.1518. PMID 1644293
- [Background] Yang MH, Chen CL, Chau GY, Chiou SH, Su CW, Chou TY, Peng WL, Wu JC. Comprehensive analysis of the independent effect of twist and snail in promoting metastasis of hepatocellular carcinoma. Hepatology. 2009 Nov;50(5):1464-74. doi: 10.1002/hep.23221. PMID 19821482
- [Background] Ogawa H, Nozawa Y, Rojanavanich V, Tsuboi R, Yoshiike T, Banno Y, Takahashi M, Nombela C, Herreros E, Garcia-Saez MI, et al. Fungal enzymes in the pathogenesis of fungal infections. J Med Vet Mycol. 1992;30 Suppl 1:189-96. doi: 10.1080/02681219280000881. No abstract available. PMID 1474443
- [Background] Calin GA, Sevignani C, Dumitru CD, Hyslop T, Noch E, Yendamuri S, Shimizu M, Rattan S, Bullrich F, Negrini M, Croce CM. Human microRNA genes are frequently located at fragile sites and genomic regions involved in cancers. Proc Natl Acad Sci U S A. 2004 Mar 2;101(9):2999-3004. doi: 10.1073/pnas.0307323101. Epub 2004 Feb 18. PMID 14973191
- [Background] Lu J, Getz G, Miska EA, Alvarez-Saavedra E, Lamb J, Peck D, Sweet-Cordero A, Ebert BL, Mak RH, Ferrando AA, Downing JR, Jacks T, Horvitz HR, Golub TR. MicroRNA expression profiles classify human cancers. Nature. 2005 Jun 9;435(7043):834-8. doi: 10.1038/nature03702. PMID 15944708
- [Background] Gregory PA, Bert AG, Paterson EL, Barry SC, Tsykin A, Farshid G, Vadas MA, Khew-Goodall Y, Goodall GJ. The miR-200 family and miR-205 regulate epithelial to mesenchymal transition by targeting ZEB1 and SIP1. Nat Cell Biol. 2008 May;10(5):593-601. doi: 10.1038/ncb1722. Epub 2008 Mar 30. PMID 18376396
- [Background] Kong W, Yang H, He L, Zhao JJ, Coppola D, Dalton WS, Cheng JQ. MicroRNA-155 is regulated by the transforming growth factor beta/Smad pathway and contributes to epithelial cell plasticity by targeting RhoA. Mol Cell Biol. 2008 Nov;28(22):6773-84. doi: 10.1128/MCB.00941-08. Epub 2008 Sep 15. PMID 18794355
- [Background] Valastyan S, Reinhardt F, Benaich N, Calogrias D, Szasz AM, Wang ZC, Brock JE, Richardson AL, Weinberg RA. A pleiotropically acting microRNA, miR-31, inhibits breast cancer metastasis. Cell. 2009 Jun 12;137(6):1032-46. doi: 10.1016/j.cell.2009.03.047. PMID 19524507 (Retraction: PMID 25879117 Cell. 2015 Apr 9;161(2):417)
- [Background] Han YC, Park CY, Bhagat G, Zhang J, Wang Y, Fan JB, Liu M, Zou Y, Weissman IL, Gu H. microRNA-29a induces aberrant self-renewal capacity in hematopoietic progenitors, biased myeloid development, and acute myeloid leukemia. J Exp Med. 2010 Mar 15;207(3):475-89. doi: 10.1084/jem.20090831. Epub 2010 Mar 8. PMID 20212066
- [Background] Gebeshuber CA, Zatloukal K, Martinez J. miR-29a suppresses tristetraprolin, which is a regulator of epithelial polarity and metastasis. EMBO Rep. 2009 Apr;10(4):400-5. doi: 10.1038/embor.2009.9. Epub 2009 Feb 27. PMID 19247375
- [Background] Xiong Y, Fang JH, Yun JP, Yang J, Zhang Y, Jia WH, Zhuang SM. Effects of microRNA-29 on apoptosis, tumorigenicity, and prognosis of hepatocellular carcinoma. Hepatology. 2010 Mar;51(3):836-45. doi: 10.1002/hep.23380. PMID 20041405
- [Background] Garzon R, Liu S, Fabbri M, Liu Z, Heaphy CE, Callegari E, Schwind S, Pang J, Yu J, Muthusamy N, Havelange V, Volinia S, Blum W, Rush LJ, Perrotti D, Andreeff M, Bloomfield CD, Byrd JC, Chan K, Wu LC, Croce CM, Marcucci G. MicroRNA-29b induces global DNA hypomethylation and tumor suppressor gene reexpression in acute myeloid leukemia by targeting directly DNMT3A and 3B and indirectly DNMT1. Blood. 2009 Jun 18;113(25):6411-8. doi: 10.1182/blood-2008-07-170589. Epub 2009 Feb 11. PMID 19211935
- [Background] Liu S, Wu LC, Pang J, Santhanam R, Schwind S, Wu YZ, Hickey CJ, Yu J, Becker H, Maharry K, Radmacher MD, Li C, Whitman SP, Mishra A, Stauffer N, Eiring AM, Briesewitz R, Baiocchi RA, Chan KK, Paschka P, Caligiuri MA, Byrd JC, Croce CM, Bloomfield CD, Perrotti D, Garzon R, Marcucci G. Sp1/NFkappaB/HDAC/miR-29b regulatory network in KIT-driven myeloid leukemia. Cancer Cell. 2010 Apr 13;17(4):333-47. doi: 10.1016/j.ccr.2010.03.008. PMID 20385359
- [Background] Mott JL, Kurita S, Cazanave SC, Bronk SF, Werneburg NW, Fernandez-Zapico ME. Transcriptional suppression of mir-29b-1/mir-29a promoter by c-Myc, hedgehog, and NF-kappaB. J Cell Biochem. 2010 Aug 1;110(5):1155-64. doi: 10.1002/jcb.22630. PMID 20564213
- [Background] Hsu DS, Lan HY, Huang CH, Tai SK, Chang SY, Tsai TL, Chang CC, Tzeng CH, Wu KJ, Kao JY, Yang MH. Regulation of excision repair cross-complementation group 1 by Snail contributes to cisplatin resistance in head and neck cancer. Clin Cancer Res. 2010 Sep 15;16(18):4561-71. doi: 10.1158/1078-0432.CCR-10-0593. Epub 2010 Sep 7. PMID 20823140
- [Background] Lin T, Ponn A, Hu X, Law BK, Lu J. Requirement of the histone demethylase LSD1 in Snai1-mediated transcriptional repression during epithelial-mesenchymal transition. Oncogene. 2010 Sep 2;29(35):4896-904. doi: 10.1038/onc.2010.234. Epub 2010 Jun 21. PMID 20562920
- [Background] Lan L, Han H, Zuo H, Chen Z, Du Y, Zhao W, Gu J, Zhang Z. Upregulation of myosin Va by Snail is involved in cancer cell migration and metastasis. Int J Cancer. 2010 Jan 1;126(1):53-64. doi: 10.1002/ijc.24641. PMID 19521958
- [Background] Martello G, Rosato A, Ferrari F, Manfrin A, Cordenonsi M, Dupont S, Enzo E, Guzzardo V, Rondina M, Spruce T, Parenti AR, Daidone MG, Bicciato S, Piccolo S. A MicroRNA targeting dicer for metastasis control. Cell. 2010 Jun 25;141(7):1195-207. doi: 10.1016/j.cell.2010.05.017. PMID 20603000
- [Background] Parra M, Verdin E. Regulatory signal transduction pathways for class IIa histone deacetylases. Curr Opin Pharmacol. 2010 Aug;10(4):454-60. doi: 10.1016/j.coph.2010.04.004. Epub 2010 May 4. PMID 20447866
- [Result] Yang MH, Chiang WC, Chou TY, Chang SY, Chen PM, Teng SC, Wu KJ. Increased NBS1 expression is a marker of aggressive head and neck cancer and overexpression of NBS1 contributes to transformation. Clin Cancer Res. 2006 Jan 15;12(2):507-15. doi: 10.1158/1078-0432.CCR-05-1231. PMID 16428493
- [Result] Yang MH, Hsu DS, Wang HW, Wang HJ, Lan HY, Yang WH, Huang CH, Kao SY, Tzeng CH, Tai SK, Chang SY, Lee OK, Wu KJ. Bmi1 is essential in Twist1-induced epithelial-mesenchymal transition. Nat Cell Biol. 2010 Oct;12(10):982-92. doi: 10.1038/ncb2099. Epub 2010 Sep 5. PMID 20818389
- [Result] Yang MH, Wu KJ. TWIST activation by hypoxia inducible factor-1 (HIF-1): implications in metastasis and development. Cell Cycle. 2008 Jul 15;7(14):2090-6. doi: 10.4161/cc.7.14.6324. Epub 2008 May 21. PMID 18635960
- [Result] Yang MH, Wu MZ, Chiou SH, Chen PM, Chang SY, Liu CJ, Teng SC, Wu KJ. Direct regulation of TWIST by HIF-1alpha promotes metastasis. Nat Cell Biol. 2008 Mar;10(3):295-305. doi: 10.1038/ncb1691. Epub 2008 Feb 24. PMID 18297062